CLINICAL TRIAL: NCT06565260
Title: Feasibility of a Community-Based Cancer Survivor Exercise and Nutrition Education Program: Effects on Self-Efficacy, Quality of Life and Functional Performance
Brief Title: Community-Based Exercise and Nutrition Training and Education Program for Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: I-3953124; NCI-2024-06518 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3953124 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (exercise/nutrition program) (Experimental): Patients participate in a supervised, community-based exercise program consisting of aerobic and resistance exercise over 45-60 minutes BIW for 12 weeks. Beginning at week 2, patients also receive nutrition education and training QW for 10 weeks. Patients also wear an activity tracker throughout the study.
  Interventions: Other: Exercise Intervention; Other: Medical Device Usage and Evaluation; Other: Nutritional Intervention; Other: Physical Performance Testing; Other: Questionnaire Administration

INTERVENTIONS:
Other: Exercise Intervention — Participate in exercise program
Other: Medical Device Usage and Evaluation — Wear an activity tracker
Other: Nutritional Intervention — Participate in nutrition program
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates whether a supervised community-based exercise and nutrition program is usable and effective for improving cancer survivors' confidence for maintaining their physical activity and nutrition. Cancer survivors often experience problems with the musculoskeletal system (bones, joints, muscles, connective tissue), the cardiopulmonary system (heart, blood vessels and lungs) and the metabolic system (how the body's cells change food into energy) following treatment. There is substantial evidence that physical activity, diet, and weight management can improve quality of life (emotional and physical well-being) and physical fitness. Information gathered from this study may help researchers determine whether participating in a community-based exercise/nutrition training and education program may improve levels of fitness, cardiovascular health, and quality of life for cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the feasibility and acceptability of a 12-week supervised community-based exercise/nutrition training and education program for cancer survivors.

SECONDARY OBJECTIVE:

I. To assess the effectiveness of a supervised exercise and nutrition training and education program by evaluating pre-post changes in exercise self-efficacy.

TERTIARY OBJECTIVE:

I. To assess changes in functional performance and quality of life (QoL).

OUTLINE:

Patients participate in a supervised, community-based exercise program consisting of aerobic and resistance exercise over 45-60 minutes twice a week (BIW) for 12 weeks. Beginning at week 2, patients also receive nutrition education and training once a week (QW) for 10 weeks. Patients also wear an activity tracker throughout the study.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Have had a previous cancer diagnosis and completed all therapy OR are a caregiver for a patient who has had a previous cancer diagnosis.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related interventions.

Exclusion Criteria:

* Have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia including atrial fibrillation (AFIB), multiple myeloma, or psychiatric illness/social situations that would limit compliance with study requirements.
* Have orthopedic or neuromuscular disorders or arthritis that preclude participation in exercise.
* Are pregnant or nursing.
* History of a stem cell transplant.
* Currently on steroids.
* Unwilling or unable to follow protocol requirements.
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-08-30 (Estimated); Study Completion 2029-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients still on study (Feasibility) | At the end of the 12 week intervention
  Feasibility will be defined as the proportion of patients still on study at the end of the 12 weeks intervention. The feasibility rate will be estimated using a 90% credible region obtained by Jeffrey's prior method. The lower bound will define a plausible lower limit for true (unobserved) feasibility rate. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies.
Percentage of patients on study after 12 weeks who complete at least 70% of intervention activities (Acceptability) | At 12 weeks
  Acceptability will be determined by measuring adherence to the intervention. The adherence rate will be considered acceptable if patients complete at least 70% of the intervention activities. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies.
Patient satisfaction (Acceptability) | Baseline to 3 months post-intervention
  Patient satisfaction will be determined through surveys. Will be summarized using the appropriate descriptive statistics and graphical summaries. Continuous variables will be summarized using the mean, median, standard deviation, and percentiles. Categorical variables will be summarized using frequencies and relative frequencies.

SECONDARY OUTCOMES:
Changes in exercise and nutrition self-efficacy | Baseline to 3 months post-intervention
  The self-reported outcomes will be summarized using the appropriate descriptive statistics. Self-reported outcomes will be compared using paired t-tests. Test assumptions will be verified graphically, and transformation or non-parametric methods (e.g., sign test) will be considered, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Ray, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States